CLINICAL TRIAL: NCT04274088
Title: The Impact of Visual Axis Position on the Optical Quality After Implantation of Multifocal Intraocular Lenses With Different Asphericity Values
Brief Title: The Clinical Importance of Angle Alpha by Multifocal Intraocular Lenses.
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Kata Mihaltz, Chief Resident, MD, PhD, Hospital Hietzing
Other Study IDs: HHietzing3
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: IOL, Cataract
Keywords: multifocal IOL, optical quality, angle alpha
MeSH Terms: conditions — Intraocular Lymphoma; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tecnis;: Patients who received the Tecnis multifocal IOL.
  Interventions: Procedure: Cataract surgery
- Diffractiva: Patients who received the Diffractiva multifocal IOL.
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Phacoemulsification surgery

SUMMARY:
Purpose: to evaluate the effect of visual axis positioning on the optical performance of the Tecnis MIOL and the Diff-aA MIOL.

DETAILED DESCRIPTION:
In this prospective, randomized comparative study 70 eyes of 35 subjects with senile cataract were implanted with the spherical aberration correcting diffractive, bifocal Tecnis ZLB00 IOL, and 60 eyes of 30 age matched subjects with the spherical aberration neutral, diffractive, bifocal Diffractiva IOL. Observation Procedure was performed 1, 3, 6 months postoperatively. Main Outcome Measures included uncorrected and corrected distance and near visual acuity, manifest refraction, ocular aberrations and visual quality metrics with 2mm and 4mm pupil, and the position of visual axis.

ELIGIBILITY:
Inclusion Criteria:

* corneal astigmatism less than 1 diopter

Exclusion Criteria:

* ocular pathology others than cataract

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients of the clinic
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 6 Month
  Schnellen VA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mihaltz K, Vecsei-Marlovits PV. The impact of visual axis position on the optical quality after implantation of multifocal intraocular lenses with different asphericity values. Graefes Arch Clin Exp Ophthalmol. 2021 Mar;259(3):673-683. doi: 10.1007/s00417-020-05052-5. Epub 2021 Jan 20. PMID 33471202